CLINICAL TRIAL: NCT01488084
Title: Comparative Evaluation of Vasomotor Function in Saphenous Veins Harvested Using Pedicled vs Conventional Technique
Brief Title: Assessing Vein Graft Properties Between Conventional & No-Touch Harvesting Technique - (PATENT SVG)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Stephen E. Fremes, Head, Division of Cardiac and Vascular Surgery, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 078-2009
Record Dates: First submitted 2011-11-07; First posted 2011-12-08 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Artery Disease
Keywords: Saphenous vein graft patency; Coronary artery bypass surgery; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pedicled "no-touch" SVG harvesting (Experimental): Saphenous vein harvested with a pedicle of surrounding fat and distension with heparinized blood at arterial pressure. No manual distention.
  Interventions: Procedure: Coronary Artery Bypass Graft Surgery
- Conventional open SVG harvesting (Active Comparator): Saphenous vein is harvested with an open technique, stripped of adventitia, and manually distended with crystalloid solution.
  Interventions: Procedure: Coronary Artery Bypass Graft Surgery; Procedure: Conventional open SVG harvesting

INTERVENTIONS:
Procedure: Coronary Artery Bypass Graft Surgery — Comparison of two techniques of saphenous vein graft harvesting for coronary artery bypass graft surgery
  Other Names: Pedicled "no-touch" saphenous vein graft harvesting; Conventional open saphenous vein graft harvesting
Procedure: Conventional open SVG harvesting — SVG harvested using conventional open technique and manually distended with crystalloid solution
  Arms: Conventional open SVG harvesting

SUMMARY:
The purpose of this study is to compare saphenous veins harvested using the atraumatic pedicled ("no-touch") technique to saphenous veins harvested using the conventional open technique in patients undergoing isolated coronary artery bypass surgery. Investigators will compare the biological structure of the saphenous veins harvested using these two techniques. There is some evidence that saphenous veins harvested using the "no-touch" technique may allow for better patency up to 8 years following bypass surgery. We may be able to detect early differences in vascular structure, observed at the time of conduit harvest.

DETAILED DESCRIPTION:
Atherosclerosis is a complex, multifactorial inflammatory disease, which is initiated largely in areas of endothelial injury, secondary to biomechanical disturbances, or systemic factors such as lipoprotein disturbances, hypertension, diabetes, and smoking (the response to injury hypothesis). Accumulating data indicate that structural and/or functional alterations in endothelial integrity play a primordial role in the development of atherosclerosis via promoting aberrant interactions between modified lipoproteins, monocyte-derived macrophages, T cells and normal cellular elements of the arterial wall inciting early plaque formation. As such, strategies, either pharmacological or mechanical in nature which reduce and/or restore endothelial homeostasis remain an important cornerstone to limit atherosclerosis.

Investigators hypothesize that saphenous veins harvested using the atraumatic pedicled ("no-touch") technique from patients undergoing isolated coronary artery bypass surgery will exhibit superior indices of vasomotor structure compared to veins harvested using the conventional open technique. We anticipate that leg healing will not be significantly altered using the "no-touch" technique.

Eligible patients will have two SVG segments harvested, one from each lower leg. One leg will have the SVG harvested in the conventional fashion and the contralateral leg will have the SVG harvested using the "no touch" technique. This will be determined by block randomization revealed at the time of skin incision. For patients with very small lower leg saphenous veins, the surgical protocol would be to then use the thigh segment instead. Patients will have Duplex scans to evaluate saphenous veins pre-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Age> 18 years and able to provide informed consent
2. Requiring isolated, primary coronary artery bypass graft surgery
3. Elective or urgent cases
4. With or without the use or cardiopulmonary bypass
5. Left ventricular ejection fraction > 20%
6. Patient require at least 2 SVG's

Exclusion Criteria:

1. Unable to give consent
2. Unable to use bilateral lower greater saphenous veins ( severe peripheral vascular disease,varicose veins, previous vein stripping, previous amputation, inadequate ultrasound appearance )
3. Pregnant women, women of child bearing age
4. Preoperative persistent atrial fibrillation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Biological Properties | Characteristics of the tissue will be reflective of the status of the tissue on the day of surgery (day 0).
  Segments of saphenous veins, approximately 5cm in length, harvested by either the conventional or no-touch technique will be employed.
  Segments will be immediately frozen in liquid nitrogen for Western blot analysis. Another 5mm segment will be used for immediate measurement of superoxide (O2-) production. Two rings, approximately 5mm in length will be frozen in Tissue Teck and another one placed in formalin (4%) and then embedded in paraffin.

SECONDARY OUTCOMES:
Leg wound Healing and Leg Functional Outcome | 12 months postoperatively
  Leg wound healing and functional outcome will be assessed in both lower legs using a quality of life measurement tool.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Fremes, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Verma S, Lovren F, Pan Y, Yanagawa B, Deb S, Karkhanis R, Quan A, Teoh H, Feder-Elituv R, Moussa F, Souza DS, Fremes SE. Pedicled no-touch saphenous vein graft harvest limits vascular smooth muscle cell activation: the PATENT saphenous vein graft study. Eur J Cardiothorac Surg. 2014 Apr;45(4):717-25. doi: 10.1093/ejcts/ezt560. Epub 2013 Dec 9. PMID 24327455